CLINICAL TRIAL: NCT04500626
Title: Multicentre Randomized Controlled Trial of Hyperbaric Versus Normobaric Oxygen Therapy for COVID-19 Patients
Brief Title: Hyperbaric Versus Normobaric Oxygen Therapy for COVID-19 Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Climate Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHRI-HBOT-001
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Covid19
Keywords: Hyperbaric oxygen therapy
MeSH Terms: conditions — COVID-19 | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBOT (Experimental): These patients will receive hyperbaric oxygen therapy (HBOT) in addition to usual treatment for COVID-19. HBOT sessions will be 75 minutes in length at a pressure of 2.0 ATA.
  Interventions: Drug: Oxygen
- Control (No Intervention): These patients will receive usual treatment for COVID-19, including oxygenation at normal atmospheric pressure (normobaric oxygenation).

INTERVENTIONS:
Drug: Oxygen — Hyperbaric oxygen therapy delivered in a monoplace or multi-place chamber. Supervised by a hyperbaric oxygen therapy physician and a chamber operator.
  Arms: HBOT

SUMMARY:
At least 1 in 6 COVID-19 patients admitted to hospital to receive extra oxygen will die of complications. In patients with COVID-19, invasive treatment such as mechanical ventilation (e.g. breathing with a machine) is associated with a 50% increased risk of death. Invasive treatments use a lot of healthcare resources in intensive care units and may lead to further deaths if patients do not have access to care.

The investigators aim to improve outcomes for COVID-19 patients by implementing hyperbaric oxygen therapy (HBOT). HBOT allows patients to breathe 100% oxygen in a special chamber at a pressure higher than sea level. It is approved by Health Canada for 14 conditions. HBOT is safe when administered by experienced teams.

There are two main causes of death in severe COVID-19 respiratory infections: (i) a decreased diffusion of oxygen from the lungs to the blood and (ii) an increased inflammatory response (also called a "cytokine storm"). HBOT leads to increased oxygen level in blood, has strong anti-inflammatory effects, and may destroy the virus responsible for COVID-19 disease. The initial experience with HBOT and COVID-19 from China, France and the United States is promising in that it prevents further worsening of the condition and need for intensive care.

The investigators propose to test the effectiveness of HBOT for COVID-19 patients who are admitted to hospital to receive extra oxygen. Using the most rigorous and innovative research methods, this Canadian-led international study will operate at 5 centers across 3 countries (Canada: Ottawa, Toronto, Edmonton; Switzerland: Geneva; UK: Rugby/London). The investigators anticipate that when treated by HBOT, COVID-19 patients needing extra oxygen to breathe will see significant health improvements as well as a decrease in complications, inflammation in the blood, need for invasive care, death, and cost of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female patients
* Age ≥18 years
* Confirmed COVID-19 positive by RT-PCR or another validated method
* Diagnosed with pneumonia requiring 21%<FIO2≤100% to maintain saturation by pulse oximetry (SpO2) ≥90%
* Able and willing to comply with study procedures and follow-up examinations contained within the written consent form

Exclusion Criteria:

* Patient clinical status felt to be incompatible with HBOT, e.g. respiratory failure requiring mechanical ventilation
* Pregnancy, determined by a serum or urine test
* Hemodynamic instability requiring vasopressors
* Inability to maintain a sitting position during treatment
* Inability to effectively understand and communicate with the hyperbaric operator, or to give consent
* Inability to spontaneously equalize ears and refusal of myringotomies
* Contraindications to HBOT (e.g. pneumothorax)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
7-level COVID Ordinal Outcome Scale | Measured on Day 7
  7-level scale based on patient's current status and need for oxygenation, also ability to resume normal activities (at higher levels). Range is 1-7. Higher number indicates better clinical outcome.

SECONDARY OUTCOMES:
Length of hospital stay | Duration of study (to Day 28)
  Measured in days
Days with oxygen supplementation | Duration of study (to Day 28)
  Number of days with oxygen supplementation
Daily oxygen flow values required to obtain saturation values ≥90%, | Duration of study (to Day 28)
  Measured in L/min
ICU admission | Duration of study (to Day 28)
  Yes/No
ICU length of stay | Duration of study (to Day 28)
  Measured in days, if applicable
Days on invasive mechanical ventilation or high flow oxygenation | Duration of study (to Day 28)
  Number of days on ventilator
Major arterial and venous thrombotic events | Duration of study (to Day 28)
  e.g. stroke, pulmonary embolism, deep vein thrombosis
Sleep quality | Duration of study (to Day 28)
  Sleep Quality Scale, measured from 0 to 10. Higher number indicates worse sleep quality: 0 = "best possible sleep", 10 = "worst possible sleep". Capelleri et. al; Health and Quality of Life Outcomes 2009: 7:54
Fatigue | Duration of study (to Day 28)
  Single-Item Fatigue Report Mark, measured from 1 to 10. Higher number indicates worse fatigue: 1 = "not at all", 10 = "extremely". van Hooff et al; J Occup Health 2007; 49:224-234.
7-level COVID Ordinal Outcome Scale | Measured on Day 28
  Same scale as the primary outcome; different timing as a secondary outcome. Range is 1-7. Higher number indicates better clinical outcome.
Mortality | Duration of study (to Day 28)
  Number of deaths
Incidence of any adverse events related to HBOT | Duration of study (to Day 28)
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Boet, MD, PhD, Principal Investigator — The Ottawa Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Rouge Valley Hyperbaric Medical Centre, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Preprint of study protocol (brief version for publication) — https://www.medrxiv.org/content/10.1101/2020.07.15.20154609v1